CLINICAL TRIAL: NCT02392767
Title: Effect of a Dietary Supplement on Endothelial Function in Volunteers With Light to Moderate Hypertension - a Randomised, Double-blind, Placebo Controlled Cross-over Study
Brief Title: Effect of L-Arginine and Pycnogenol on Light to Moderate Hypertension and Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Loges & Co. GmbH (Industry)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BTS815/14
Record Dates: First submitted 2014-11-14; First posted 2015-03-19 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-03

CONDITIONS: Endothelial Dysfunction; Hyperhomocysteinemia; Hypertension Grade I, Subgroup "Borderline" (WHO)
Keywords: L-Arginine; Pycnogenol; vitamin K2; vitamin B; endothelial function; hypertension; Homocystein >10
MeSH Terms: conditions — Hyperhomocysteinemia; Hypertension | interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum (Active Comparator): 2 times 2 tablets a day for 4 weeks.
  Interventions: Dietary Supplement: Verum
- Placebo (Placebo Comparator): 2 times 2 tablets a day which cornstarch. Tablets look identical like verum tablets.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Verum — 2400 mg L-arginine, 80 mg Pycnogenol, 45µg vitamine K2, 10 mg R (+) alpha lipoic acid, 8 mg vitamine B6, 500 µg vitamine B12, and 600 mg folic acid.
  Arms: Verum
Dietary Supplement: Placebo — corn starch
  Arms: Placebo

SUMMARY:
The effect of a combination product (Verum ) with L-arginine, Pycnogenol, vitamin K2, R-(+)-alpha-lipoic acid and vitamins B6, B12 and folic acid is investigated in a double blind placebo-controlled cross-over study. Volunteers with hypertension and hyperhomocysteinemia are randomly assigned to the dietary supplement or placebo.

DETAILED DESCRIPTION:
25 patients were included in the trial. Intervention period was 4 weeks with 2 months wash out phase. The screening visit of all volunteers before study start included volunteer information, signature of informed consent, anamnesis, medical history, ECG and blood routine analysis.

Efficacy parameters were measured at visit 1, 2, 3, and 4. Endothelial function and postprandial endothelial Reaction was tested using EndoPAT (validated diagnosis tool). Blood pressure was measured by volunteers over a period of 7 days before each visit. As additional parameters homocysteine and ADMA (assymmetric dimethyl arginine) were determed. For safety evaluation AEs (Adverse Events), CC (compliance control), tolerability, blood routine parameters and vital signs were assessed.

ELIGIBILITY:
Inclusion Criteria:

* borderline blood pressure (systolic 130-149)
* homocystein level >10µmol/l

Exclusion Criteria:

e.g.

* BMI <20kg/m2 and >32kg/m2
* use of antihypertensives, anticoagulants, and statins
* cardiovascular diseases e.g. stroke, myocardial infarction
* use of L-arginine and other dietary supplements

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Goyvaerts, Dr., Study Chair — medical advisor
Locations (1):
- BioTeSys, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] Reule CA, Goyvaerts B, Schoen C. Effects of an L-arginine-based multi ingredient product on endothelial function in subjects with mild to moderate hypertension and hyperhomocysteinemia - a randomized, double-blind, placebo-controlled, cross-over trial. BMC Complement Altern Med. 2017 Feb 2;17(1):92. doi: 10.1186/s12906-017-1603-9. PMID 28153005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cross-over study
Groups:
- First Verum, Then Placebo: 2 times a day 2 verum tablets for 4 weeks. 8 weeks wash out. Then 2 times a day 2 placebo tablets for 4 weeks.
- First Placebo, Then Verum: 2 times a day 2 placebo tablets for 4 weeks. 8 weeks wash out. Then 2 times a day 2 verum tablets for 4 weeks.
Period: Overall Study
Arm/Group | First Verum, Then Placebo | First Placebo, Then Verum
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First Verum, Then Placebo | First Placebo, Then Verum | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  Germany | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Endothelial Function Between the Visit at Start of Supplementation Phase and the Visit on the Final Day of the 4 Week Supplementation Phase (Delta "lnRHI")
Description: Endothelial function was determined with the EndoPAT™ method (non-invasive Peripheral Aterial Tonometry) using a reactive hyperemia procedure. The outcome measure is the change in endothelial function between the visit at start of the supplementation phase and the visit on the final day of the 4 week supplementation phase. The endothelial function is determined as the natural log of the Reactive Hyperemia Index ("lnRHI") which is the post-to-pre occlusion peripheral arterial tonometry signal ratio in the occluded side, relative to the same ratio in the control side, corrected for baseline vascular tone of the occluded side.
  Normal lnRHI > 0.51, Abnormal lnRHI < 0.51
Time Frame: Intervention period of 4 weeks
Measure: Mean (95% Confidence Interval); unit: Delta lnRHI [Index]
Groups:
- Placebo: 2 times 2 tablets a day for 4 weeks.
  Placebo: corn starch
Arm/Group | Verum | Placebo
Number analyzed (Participants) | 25 | 25
Delta lnRHI [Index] | 0.070 [-0.065 to 0.205] | -0.052 [-0.163 to 0.060]

2. Secondary Outcome: Mean of Blood Pressure Measured Daily at the Last 7 Days of the 4 Week Intervention Period.
Description: The mean of daily systolic and diastolic blood pressure measured daily at the last 7 days of the 4 week intervention period. Measurements were performed by subjects at home and were taken on the left arm, after at least 10 minutes of rest, in a sitting position.
Time Frame: Intervention period of 4 weeks
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Placebo: 2 times 2 tablets a day for 4 weeks
  Placebo: corn starch
Arm/Group | Verum | Placebo
Number analyzed (Participants) | 25 | 25
mmHg
  systolic reading | 132.8 [129.1 to 136.6] | 133.2 [130.4 to 136.1]
  diastolic reading | 82.2 [79.8 to 84.6] | 83.5 [81.7 to 85.3]

3. Secondary Outcome: Homocystein Level Determined on the Final Day of the 4 Week Intervention Period.
Description: Homocystein level in µmol/l was determined on the final day of the 4 week intervention period.
  The first supplementation period started at visit one and lasted for 4 weeks. It was followed by a wash out phase of 8 weeks and subsequently by a second supplementation phase of 4 weeks (cross-over design)
Time Frame: After intervention period of 4 weeks
Measure: Mean (95% Confidence Interval); unit: μmol/l
Arm/Group | Verum | Placebo
Number analyzed (Participants) | 25 | 25
μmol/l | 9.10 [8.30 to 9.90] | 11.95 [11.19 to 12.72]

4. Secondary Outcome: Asymmetric Dimethyl Arginine (ADMA) Level Determined on the Final Day of the 4 Week Intervention Period.
Description: ADMA (asymmetric dimethyl arginine) was determined on the final day of the 4 week intervention period. Samples were analyzed batch wise using an enzymatic test
Time Frame: After intervention period of 4 weeks
Measure: Mean (95% Confidence Interval); unit: µmol/l
Arm/Group | Verum | Placebo
Number analyzed (Participants) | 25 | 25
µmol/l | 0.638 [0.594 to 0.682] | 0.632 [0.596 to 0.668]

5. Secondary Outcome: Glycated Hemoglobin (HbA1c) Determined on the Final Day of the 4 Week Intervention Period.
Description: Glycated hemoglobin (HbA1c) as percentage of total hemoglobin was determined on the final day of the 4 week intervention period.
Time Frame: After intervention period of 4 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of total hemoglobin
Arm/Group | Verum | Placebo
Number analyzed (Participants) | 25 | 25
percentage of total hemoglobin | 5.37 [5.20 to 5.54] | 5.34 [5.19 to 5.50]

6. Other Pre Specified Outcome: Change in Prothrombin Time Between the Visit at Start of Supplementation Phase and the Visit on the Final Day of the 4 Week Supplementation Phase
Description: Prothrombin Time was assessed at the visit at start of the supplementation phase and the visit at the end of the 4 week supplementation phase. Blood coagulability is expressed in units of Quick value. In this case, the measured prothrombin time is expressed in relation to the coagulation time of a healthy person. The value obtained is the "percentage of the standard Quick value". In a person not receiving oral anticoagulation the "normal" Quick value is between 70 and 100%. The longer the patient's coagulation time, the lower the Quick value
Time Frame: Intervention period of 4 weeks
Measure: Mean (95% Confidence Interval); unit: Percentage of the standard Quick value
Arm/Group | Verum | Placebo
Number analyzed (Participants) | 25 | 25
Percentage of the standard Quick value | 2.00 [-0.54 to 4.54] | 1.50 [-1.31 to 4.31]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Verum | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 9/25 | 12/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verum (N=25) | Placebo (N=25)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
cold (Infections and infestations) | 2 (2) | 1 (1) — common cold
headache (Nervous system disorders) | 2 (2) | 2 (3)
malaise (Gastrointestinal disorders) | 0 (0) | 1 (1) — stomach upset with diarrhoea
nasal mucosa disorder (Surgical and medical procedures) | 0 (0) | 1 (1)
loose stools (Gastrointestinal disorders) | 0 (0) | 1 (1)
herpes NOS (Infections and infestations) | 0 (0) | 1 (1)
febrile infection (Infections and infestations) | 0 (0) | 3 (3)
gastrointestinal infection (Gastrointestinal disorders) | 0 (0) | 1 (1)
lumbago (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
generalized aching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — after gardening
skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
bladder infection (Renal and urinary disorders) | 1 (1) | 0 (0)
cycling accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No